CLINICAL TRIAL: NCT04018352
Title: Assessment of Variations of The Number of Roots &Amp; Root Canal Configurations of Maxillary Premolars and Their Relation to the Floor of the Maxillary Sinus in a Sample of Egyptian Population Using CBCT: An Observational Cross-Sectional Study
Brief Title: Assessment of Variations of The Number of Roots &Amp; Root Canal Configurations of Maxillary Premolars and Their Relation to the Floor of the Maxillary Sinus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Khairy Morsy, Principal Investigator, Cairo University
Other Study IDs: ORAD7-1-1
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Root Canal Configurations of Permanent Maxillary Premolars

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of Variations of The Number of Roots & Root Canal Configurations of Permanent Maxillary Premolars and their Relation to the Floor of the Maxillary sinus

DETAILED DESCRIPTION:
Assessment of Variations of The Number of Roots & Root Canal Configurations of Permanent Maxillary Premolars and their Relation to the Floor of the Maxillary sinus in a Sample of Egyptian Population using CBCT: An Observational Cross-Sectional Study

ELIGIBILITY:
Inclusion Criteria:

* Fully maturated and erupted maxillary permanent premolars of Egyptian patients, males or females.
* Intact maxillary premolars' roots without fractures or cracks.
* Maxillary Premolars without posts or previous root canal treatment.
* CBCT scans of different fields of view could be included as long as it shows maxillary premolars.
* CBCT scans of 0.2 mm voxel resolution {the maximum voxel size accepted for endodontic imaging}

Exclusion Criteria:

* Maxillary premolars with:

Developmental anomalies. External or internal root resorption. Root canal calcification. Previous root canal treatment Post restorations. Root caries especially reaching the bifurcation area.

* Evidence of apicectomy or periapical surgery
* CBCT images of poor quality or artifacts interfering with the assessment of the root canals.

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian Population
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2019-07-30 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of roots maxillary premolars | up to 2020
  Detection of number of maxillary roots in Egyptian population

SECONDARY OUTCOMES:
Assessment of the relationship between maxillary premolars roots and the maxillary sinus floor | up to 2020
  Recording of the relationship between maxillary premolars roots and the maxillary sinus floor

OTHER OUTCOMES:
Number of root canals | up to 2020
  Counting the number of root canals
Root canals configuration | up to 2020
  Detection of root canals configuration